CLINICAL TRIAL: NCT01315405
Title: Do Facial Expression Recognition Disorder and Mirror Neurons Subtend Apathy in Parkinson's Disease?
Brief Title: Facial Expression Recognition and Mirror Neurons in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0090
Record Dates: First submitted 2011-02-28; First posted 2011-03-15 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Parkinson's Disease
Keywords: Emotional facial expression; Apathy; Mirror neurons
MeSH Terms: conditions — Parkinson Disease; Lethargy

INTERVENTIONS:
Behavioral: Emotional facial expression recognition tests — 20 patients with an Idiopathic Parkinson's disease
  + 20 paired healthy volunteers (on sex, age, and education)
  After inclusion, patients are evaluated two times: they are studied without medication (MED OFF) and with medication (STIM ON) in a randomized order. The 2 evaluations should be spaced out 15 days to one month (J0 and J+15d)
  Healthy subjects have only one visit J0 (inclusion and emotional facial expression recognition tests are made at the same time)

SUMMARY:
After few years of evolution, patients with Parkinson's disease may develop apathy, with different degrees of severity. Apathy is characterized by a loss of interest for the others and for activities. The lack of social interactions in these patients may be due to an impairment in decoding emotional facial expression. Indeed, facial expression recognition, which is necessary to understand other's emotional state, requires a subclinical facial mimicking of the expression observed. Yet, one of the clinical signs of PD is amimia.

This study aims to determinate if there is a facial mimicry disorder in PD ( Parkinson's disease )patients with emotional facial expression (EFE) recognition impairment, compared to healthy control subjects. We also want to know if this facial mimicry disorder is primary (subtended by facial mobility impairment, that is to say amimia) or secondary (related to the mirror neuron systems that allows us to activate similar neural networks when observing and feeling a specific emotion)

DETAILED DESCRIPTION:
20 patients with an Idiopathic Parkinson's disease

+ 20 paired healthy volunteers (on sex, age, and education)

After inclusion, patients are evaluated two times: they are studied without medication (MED OFF) and with medication (STIM ON) in a randomized order. The 2 evaluations should be spaced out 15 days to one month (J0 and J+15d)

Healthy subjects have only one visit J0 (inclusion and emotional facial expression recognition tests are made at the same time)

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease according to UKPDSBB criteria - Men or women aged between 18 to 75 years
* Free from any visio-perceptive disorder (visual acuity and Vitec)
* Affiliated to National Health system
* Having given their informed consent

  --Healthy controls
* Men or women aged between 18 to 75 years
* Free from any visio-perceptive disorder (visual acuity and Vitec)
* Affiliated to National Health system
* Having given their informed consent

Exclusion Criteria:

* With dementia or with significant dysexecutive disorder (MMS <24, MATTIS< 130)
* With fluctuations (<5 Levodopa intakes / day)
* With severe depression (BDI > 27)
* With psychiatric comorbidities (hallucinations, psychos) evaluated with l'Unified Parkinson's disease Rating Scale part I (UPDRS part I =0)
* With faces processing disorder (Benton < 39)
* Pregnant
* Treatment with deep brain stimulation
* Under guardianship
* In excluding period for another study

  --Healthy controls
* Suffering of neurological or psychiatric evolutive condition
* With severe depression (BDI > 27)
* With faces processing disorder (Benton < 39)
* Pregnant
* In excluding period for another study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of facial electromyographic activity during emotional facial expression recognition tests | at J0 and at J+15 days

SECONDARY OUTCOMES:
Measurement of facial electromyographic activity during voluntary facial mimicking | at J0 and at J+15days
Measurement of facial electromyographic activity during emotional movies viewing | Made at J0 and at J+15days
Measurement of Empathy (Baron-Cohen), Apathy (Starkstein) | Made at J0 and at J+15days
Measurement of the effect of Levodopa on these parameters | Made at J0 and at J+15days

CONTACTS AND LOCATIONS:
Overall Officials: Ana MARQUES, PH, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France